CLINICAL TRIAL: NCT02866305
Title: Thoracoscopic Treatment of Primary Pneumothorax - A National Randomised Controlled Trial
Brief Title: Study Designed to Optimize the Treatment of Primary Pneumothorax
Acronym: TOPP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Medical Association (Other); Danmarks Lungeforening (Other)
Responsible Party: Principal Investigator, Winnie Hedevang Olesen, MD and Principal investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOPP2009
Record Dates: First submitted 2010-08-09; First posted 2016-08-15 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Primary Spontaneous Pneumothorax; Pleural Disease
Keywords: primary spontaneous pneumothorax; epidemiology; genetics; risk factors
MeSH Terms: conditions — Pneumothorax; Pleural Diseases | interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HRCT with bullae, treatment conservative (Experimental): Patients undergo High-resolution CT scan, and significant bullae are identified (i.e. > 1 cm). Afterwards randomised to conservative treatment with conventional chest-tube drainage.
  Interventions: Procedure: Chest tube insertion; Radiation: High-resolution Computer Tomography
- HRCT no bullae, treatment conservative (Experimental): Patients undergo High-resolution CT scan, and no significant bullae are identified (i.e. > 1 cm). Afterwards randomised to conservative treatment with conventional chest-tube drainage.
  Interventions: Procedure: Chest tube insertion; Radiation: High-resolution Computer Tomography
- HRCT with bullae, treatment VATS. (Experimental): Patients undergo High-resolution CT scan, and significant bullae are identified (i.e. > 1 cm). Afterwards randomised to active treatment with VATS bullectomy and mechanical pleurodesis.
  Interventions: Procedure: VATS bullectomy and mechanical pleuradesis.; Procedure: Chest tube insertion; Drug: Epidural; Radiation: High-resolution Computer Tomography
- HRCT no bullae, treatment VATS. (Experimental): Patients undergo High-resolution CT scan, and no significant bullae are identified (i.e. > 1 cm). Afterwards randomised to active treatment with VATS bullectomy and mechanical pleurodesis.
  Interventions: Procedure: VATS bullectomy and mechanical pleuradesis.; Procedure: Chest tube insertion; Drug: Epidural; Radiation: High-resolution Computer Tomography

INTERVENTIONS:
Procedure: VATS bullectomy and mechanical pleuradesis. — Thoracoscopic bullectomy is performed on all visible bullae, alternatively is no visible bullae, the apex is resected. Then mechanical pleuradesis is performed.
  Arms: HRCT no bullae, treatment VATS.; HRCT with bullae, treatment VATS.
Procedure: Chest tube insertion — Conventional chest tube insertion.
Drug: Epidural — All surgical participants received an epidural prior to the procedure.The epidural was removed simultaneous with the the chest tube.
  Other Names: Pain- catheter
  Arms: HRCT no bullae, treatment VATS.; HRCT with bullae, treatment VATS.
Radiation: High-resolution Computer Tomography — All participants included in this study had a HRCT performed.

SUMMARY:
Knowledge about incidence, risk factors and genetic predispositions of primary spontaneous pneumothorax in young adults is very limited, and treatment has also been controversial.The Aim of this study is to optimize the treatment, estimate the actual incidence, and identify possible risk factors including genetic predispositions.

DETAILED DESCRIPTION:
* Background Knowledge about incidence, risk factors and genetic predispositions of primary spontaneous pneumothorax in young adults is very limited, and treatment has also been controversial. Typically, the first incidence is treated conservatively with simple chest tube drainage and only if the disease reoccurs is surgery considered. However, conventional treatment may be associated with increased morbidity, prolonged hospitalization and many young adults are concerned about the high recurrence of this disease. The latter has been reported in as many as 25-35% of patients. Because spontaneous pneumothorax in young adults usually is associated with apical blebs, the investigators hypothesized that primary surgery (Video-Assisted Thoracoscopic Surgery = VATS) with resection of such blebs at the time of the first episode of pneumothorax might be an effective first line treatment associated with lower morbidity and shorter hospital stays, and a definite decline in recurrence rate.
* Method From July 2009 the investigators conducted a nationwide study , where 300 consecutive patients admitted to a Danish hospital with primary spontaneous pneumothorax undergo a high resolution CT of the thorax. Based upon the CT the patients are randomised to conventional conservative treatment (chest tube drainage) or primary VATS with bleb resection and mechanical pleurodesis.

Participants are followed for ten years. The primary endpoint is ipsilateral recurrence of pneumothorax. Secondary endpoints are length of hospitalization, duration of chest tube drainage and miscellaneous complications.

Simultaneously, a research biobank containing blood samples and pulmonary tissue is created for future studies of biomarkers and possible genetic causes.

Finally, the investigators are conducting a national epidemiological study, where the incidence in the Danish population is investigated.

*Perspective This study contributes new knowledge on incidence, genetics and best treatment of primary spontaneous pneumothorax in young adults which will have an impact on the future strategy of both understanding and treatment of this disease on a global level.

ELIGIBILITY:
Inclusion Criteria:

* First incidence of primary spontaneous pneumothorax.
* Age between 18 and 40.
* No known preexisting pulmonary disease.
* Patient must accept randomization.
* Able to read and understand information regarding the study.
* The condition must require treatment with a chest-tube.

Exclusion Criteria:

* Age above 40.
* Previously pulmonary og cardiac surgery.
* Pregnant or breastfeeding.
* Patients who do not tolerate anesthetics.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-03; Primary Completion 2017-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to ipsilateral recurrence | 10 years
  All participants are followed 10 years from the initial discharge via Questionnaires

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 10 years
Length of hospital stay | up to 10 years
  Length of initial hospital stay
Pain according to NRS scale reported at discharge, at 4 weeks, 1 year, 5 years and 10 years. | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Hedevang Olesen, ph.d.student, Study Director — Research Unit at the Cardiothoracic Department at the University Hospital of Odense.; Peter Bjørn Licht, Professor MD, Principal Investigator — Research Unit at the Cardiothoracic Department at the University Hospital of Odense
Locations (3):
- Denmark (3):
  - Research Unit at the Cardiothoracic Department at the University Hospital of Skejby, Aarhus, Central Jutland
  - Research Unit at the cardiothoracic departement at the University Hospital of Odense, Odense, Fyn
  - Research Unit at the Cardiothoracic Department af Ålborg Hospital, Aalborg, North Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olesen WH, Katballe N, Sindby JE, Titlestad IL, Andersen PE, Lindahl-Jacobsen R, Licht PB. Surgical treatment versus conventional chest tube drainage in primary spontaneous pneumothorax: a randomized controlled trial. Eur J Cardiothorac Surg. 2018 Jul 1;54(1):113-121. doi: 10.1093/ejcts/ezy003. PMID 29509892